CLINICAL TRIAL: NCT02641067
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MK-1439 (Doravirine) in Subjects With Severe Renal Impairment
Brief Title: A Study Evaluating the Pharmacokinetics of Doravirine (MK-1439) in Participants With Severe Renal Impairment (MK-1439-051)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1439-051; MK-1439-051 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Severe Renal Impairment (Experimental): Participants with severe renal impairment receive a single oral dose of 100 mg doravirine
  Interventions: Drug: Doravirine
- Healthy Matched Control (Experimental): Healthy participants matched for age and weight receive a single oral dose of 100 mg doravirine
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — Following an overnight fast, a single coated tablet of 100 mg doravirine will be administered orally
  Other Names: MK-1439, PIFELTRO

SUMMARY:
This study will evaluate the effect of severe renal impairment on the pharmacokinetics of doravirine.

ELIGIBILITY:
Inclusion Criteria:

* is a non-smoker or moderate smoker
* has a body mass index (BMI) ≥ 18.5 and ≤ 40.0 kg/m^2
* other than renal impairment, participant is judged to be in good health based on medical history, physical examination, vital signs, and laboratory safety tests
* female informed of the risks of pregnancy, agree not to become pregnant while participating in this study. Female of childbearing potential must either be sexually inactive for 14 days prior to dosing and throughout the study, or uses one acceptable birth control method
* female of non-childbearing potential must have undergone sterilization procedures at least 6 months prior to dosing.
* Participants with severe renal impairment only: has baseline estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2

Exclusion Criteria:

* is mentally or legally incapacitated or has significant emotional problems
* has a history or presence of clinically significant medical or psychiatric condition or disease
* has history or presence of alcoholism or drug abuse within the past 2 years
* has history or presence of hypersensitivity or idiosyncratic reaction to the study drug, any inactive ingredients, or related compounds
* has history or presence of renal artery stenosis
* has had a renal transplant or nephrectomy
* has rapidly fluctuating renal function as determined by historical measurements
* female is pregnant or lactating
* has positive results for the urine or saliva drug and urine or breath alcohol screen at screening or check-in
* has positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)
* is unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to dosing and throughout the study. Certain medications including those to treat kidney disease will be permitted. Other medications may be permitted following consultation with the Sponsor Clinical Monitor.
* is unable to refrain from or anticipates the use of inducers of cytochrome P450 3A (CYP3A) or permeability glycoprotein (P-gp) transporters for at least 28 days prior to dosing and throughout the study.
* has been on a diet incompatible with the on-study diet, within 28 days prior to dosing, and throughout the study
* has donated blood or had significant blood loss within 56 days prior to dosing
* has donated plasma within 7 days prior to dosing
* has participated in another clinical trial within 28 days prior to dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2016-05-14 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ankrom W, Yee KL, Sanchez RI, Adedoyin A, Fan L, Marbury T, Preston RA, Iwamoto M, Khalilieh SG. Severe Renal Impairment Has Minimal Impact on Doravirine Pharmacokinetics. Antimicrob Agents Chemother. 2018 Jul 27;62(8):e00326-18. doi: 10.1128/AAC.00326-18. Print 2018 Aug. PMID 29891610

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe Renal Impairment: Participants with severe renal impairment received a single oral dose of 100 mg doravirine
- Healthy Matched Controls: Healthy participants matched for age and weight received a single oral dose of 100 mg doravirine
Period: Overall Study
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impairment | Healthy Matched Controls | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Customized [Count of Participants; unit: Participants]
  19 to 49 years | 0 | 0 | 0
  50 to 59 years | 4 | 4 | 8
  60 to 69 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 5 | 11
Body Weight [Mean (Standard Deviation); unit: Kilogram] | 90.86 (17.409) | 90.93 (6.086) | 90.89 (12.599)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 Hours to Infinity (AUC0-∞) of Doravirine
Description: Blood was collected for the determination of plasma doravirine using a liquid chromatographic tandem mass spectrometric method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 12, 24, 48, 72 hours post-dose for all participants; and 96 hours post-dose for participants with severe renal impairment
Population: All participants who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: μM•hr
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
μM•hr | 64.5 [47.4 to 87.8] | 45.1 [33.2 to 61.4]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy Matched Controls; Test type: Other; Geometric mean ratio = 1.43, 90% CI 2-sided [1.00 to 2.04]

2. Primary Outcome: Plasma Concentration of Doravirine at 24 Hours Postdose (C24)
Description: as for outcome 1
Time Frame: 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
nM | 943 [710 to 1250] | 684 [515 to 908]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy Matched Controls; Test type: Other; Geometric mean ratio = 1.38, 90% CI 2-sided [0.99 to 1.92]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Doravirine
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: nM
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
nM | 1580 [1210 to 2080] | 1900 [1450 to 2500]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy Matched Controls; Test type: Other; Geometric mean ratio = 0.83, 90% CI 2-sided [0.61 to 1.15]

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 Hours to the Time of Last Quantifiable Sample of Doravirine (AUC 0-last)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM•hr
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
μM•hr | 60.5 (56.3) | 41.0 (29.9)

5. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Doravirine
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
Hours | 2.00 [0.50 to 4.00] | 1.50 [0.50 to 6.00]

6. Primary Outcome: Apparent Terminal Half-life (t1/2) of Plasma Doravirine
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
Hours | 25.02 (36.4) | 16.69 (26.1)

7. Primary Outcome: Apparent Clearance of Plasma Doravirine After Extravascular Administration (CL/F)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
Liter/hour | 3.53 (63.9) | 5.38 (32.8)

8. Primary Outcome: Apparent Volume of Distribution of Plasma Doravirine During the Terminal Phase (Vz/F)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Severe Renal Impairment | Healthy Matched Controls
Number analyzed (Participants) | 8 | 8
Liters | 127 (40.9) | 129 (28.3)

ADVERSE EVENTS:
Time Frame: Up to 14 days after drug administration
Description: The population analyzed consisted of all participants who received at least 1 dose of study treatment.
Groups:
- Healthy Matched Control: Healthy participants matched for age and weight received a single oral dose of 100 mg doravirine
Arm/Group | Severe Renal Impairment | Healthy Matched Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Renal Impairment (N=8) | Healthy Matched Control (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's policy on authorship is consistent with the requirements outlined in the ICH-Good Clinical Practice guidelines. In summary, authorship should reflect significant contribution to the design and conduct of the trial, performance or interpretation of the analysis, and/or writing of the manuscript.